CLINICAL TRIAL: NCT04838938
Title: Personalized Medicine in Patients With Infective Endocarditis
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Responsible Party: Sponsor
Other Study IDs: FINBA_critlab_4
Record Dates: First submitted 2021-03-26; First posted 2021-04-09 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Infective Endocarditis; Response, Acute Phase; Treatment
MeSH Terms: conditions — Endocarditis; Acute-Phase Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Samples with DNA for the study of the host's sub phenotypes Plasma and heart valves to make a metagenomic sequencing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hypothesis underlying this work is the identification of different sub phenotypes of patients with infective endocarditis through the study of the host's response to infection.

Furthemore, metagenomic sequencing may be a helpful supplement to IE diagnostic, especially when conventional tests fail to yield a diagnosis.

DETAILED DESCRIPTION:
Infective endocarditis is a life-threatening infection of heart valves and adjacent structures characterized by vegetations on valves and other endocardial surfaces, with tissue destruction and risk of embolization.

The clinical variability, including the heterogeneous response to infection and the different antibiotic treatments make the identification of the underlying pathogens of infective endocarditis (IE) is critical for precision therapy. Virulence factors mediate tissue adherence, host infiltration, immune resistance/evasion, and dynamic stress responses and confer enhanced pathogen survival, proliferation, and host invasion in animal models of infective endocarditis.

To identify the microorganism and simultaneously considered the response of the host to the infection could improve the management of the infective endocarditis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active infective endocarditis according to the modified Duke criteria.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an active infective endocarditis
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
To characterize a cohort of patients diagnosed with infective endocarditis | 2 year
  Clinical, microbiological and echocardiographic description of patients with infective endocarditis.

SECONDARY OUTCOMES:
Identification of the underlying pathogens of infective endocarditis (IE) | 2 year
  We will employ next-generation sequencing for pathogens and antimicrobial resistance detection in IE patients.
Host response classification for infective endocarditis (IE) | 2 year
  Differential baseline expression of some genes may indicate resilience to infection.
Host response predictors of sepsis outcomes | 2 year
  We will develop and use advanced bioinformatic, metabolomic, proteomic and mRNA sequencing technologies to identify specific changes, or biomarkers, in patient blood samples that predict outcome in sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Muñiz Albaiceta, MD, PhD, Study Director — HUCA-FINBA, Universidad de Oviedo
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Yes
All datasets underlying the study are available upon request to the study principal investigator.
  All of the individual participant data collected during the trial, informed consent forms, study protocol, statistical analysis plan and raw data, are available under reasonable request, and after deindentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting 3 month after publication
Access Criteria: Principal investigator will review requests of data to be provided.